CLINICAL TRIAL: NCT05583136
Title: Restoring Neural Oscillatory Communication Between Dorsal and Ventral Visual Streams in Developmental Dyslexia
Brief Title: Restoring Neural Oscillatory Communication in Developmental Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Luca Ronconi, Professor, IRCCS Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NeOsReDy-01
Record Dates: First submitted 2022-10-07; First posted 2022-10-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-10

CONDITIONS: Developmental Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group DD1 (Experimental): tACS + visuo-attentional training
  Interventions: Device: Parietal tACS combined with visuo-attentional training
- Group DD2 (Active Comparator): Sham (placebo) tACS + visuo-attentional training
  Interventions: Device: Sham (placebo) tACS combined with visuo-attentional training
- Group DD3 (Active Comparator): Sham (placebo) tACS + phonics training
  Interventions: Device: Sham (placebo) tACS combined with phonics training

INTERVENTIONS:
Device: Parietal tACS combined with visuo-attentional training — Parietal tACS combined with visuo-attentional training
  Arms: Group DD1
Device: Sham (placebo) tACS combined with visuo-attentional training — Sham (placebo) tACS combined with visuo-attentional training
  Arms: Group DD2
Device: Sham (placebo) tACS combined with phonics training — Sham (placebo) tACS combined with phonics training
  Arms: Group DD3

SUMMARY:
Developmental dyslexia (DD) is a multifactorial disorder that hampers the education of about 10% of individuals across cultures and is associated to both phonological and visual deficits. The latter have been linked to a deficit in the magnocellular-dorsal (M-D) visual stream, that has a critical role in guiding the activity of ventral visual stream areas where letters identity is extracted. Here, we will test the efficacy of transcranial alternate current stimulation (tACS) of the M-D stream combined with reading trainings in adult participants with DD, assessing the neurophysiological underpinnings of these new trainings with EEG and fMRI/DTI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age between 18 and 35)
* Official Diagnosis of Developmental Dyslexia (DD)
* Normal or corrected-to-normal vision and hearing
* Normal motor skills

Exclusion Criteria:

* Participants that cannot sign the consent form
* Participants unable to read or understand and correctly complete the procedures foreseen by the study
* Participants with a diagnosis or personal history of epilepsy or patients with a positive family history of epilepsy
* Pregnant or breastfeeding patients
* Participants with major psychiatric or neurological disorders and/or currently in psychopharmacological treatments.
* Participants with metal implants in the brain, pacemakers, brain stimulators, cochlear implants.
* Participants with claustrophobia (only for fMRI)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Reading score | Pre-training, 1-7 days post-training, follow-up at 1 and 6 months
  Text, word and pseudowords reading score

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Ronconi, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided